CLINICAL TRIAL: NCT00292253
Title: A Randomized, Multicenter, Parallel Group, Open-label Study Comparing the Tolerability of Rebif® Injection With and Without the Use of Rebiject™Mini in Relapsing Remitting MS Patients
Brief Title: Tolerability of Rebif® Injection With and Without the Use of Rebiject™Mini in Relapsing-Remitting Multiple Sclerosis Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22982
Record Dates: First submitted 2006-02-13; First posted 2006-02-15 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: Multiple Sclerosis, Relapsing-remitting
Keywords: MS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

ARMS (2):
- Rebif® with Rebiject™Mini (Experimental)
  Interventions: Device: Rebif® via Rebiject™Mini
- Rebif® without Rebiject™Mini (Active Comparator)
  Interventions: Device: Rebif® via manual injections

INTERVENTIONS:
Device: Rebif® via Rebiject™Mini — Rebif® will be administered subcutaneously at a dose 44 mcg three times a week with Rebiject™Mini, an auto-injection device for 3 months.
  Arms: Rebif® with Rebiject™Mini
Device: Rebif® via manual injections — Rebif® will be administered subcutaneously at a dose 44 mcg three times a week with manual injections for 3 months.
  Arms: Rebif® without Rebiject™Mini

SUMMARY:
This is a randomized, multicenter, parallel-group, open-label study comparing the tolerability of Rebif® injections (44 microgram [mcg] administered subcutaneously three times a week) with and without Rebiject™Mini, an auto-injection device in relapsing-remitting multiple sclerosis (MS) subjects. Subjects will be randomly assigned to either one of the two Rebif® groups in a 1:1 ratio on Study Day 1 stratified by center. Subjects will receive a minimum of 3 months of treatment with Rebif® 44 mcg three times a week and will be asked to assess their injection site reactions on a weekly basis. Clinic visit will occur at 1 and 3 months after the initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age
* Has relapsing-remitting MS
* Are willing and able to comply with the protocol for the duration of the study

Exclusion Criteria:

* Has significant leukopenia/lymphopenia (white blood cell count less than (<) 0.5 times the lower limit of normal)
* Has elevated liver function tests (aspartate aminotransferase [AST], Alanine transaminase [ALT], or alkaline phosphatase greater than (>) 2 times the upper limit of normal or total bilirubin > 1.5 times the upper limit of normal)
* Has an allergy to human serum albumin or mannitol
* Had treatment with an investigational product or procedure within 3 months
* Has the presence of systemic disease or abnormal laboratory findings that might interfere with subject safety, compliance or evaluation of the condition under study
* Has concomitant use of Avonex®, Betaseron®, Copaxone®, or Novantrone®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1883 (Actual)
Dates: Start 2001-01; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with moderate to severe (Grade 3-5) injection site reactions based on physician assessment | Month 3

SECONDARY OUTCOMES:
Number of subjects with any injection site reactions based on physician assessment | Month 3
Percentage of moderate to severe (Grade 3-5) injection site reactions reported per subject based on subject reports | Baseline up to Month 3
Percentage of injection site reactions reported per subject based on subject reports | Baseline up to Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Maria Lopez-Bresnahan, M.D., Study Director — Merck Serono International SA

REFERENCES:
- [Result] Mikol D, Lopez-Bresnahan M, Taraskiewicz S, Chang P, Rangnow J; Rebiject Study Group. A randomized, multicentre, open-label, parallel-group trial of the tolerability of interferon beta-1a (Rebif) administered by autoinjection or manual injection in relapsing-remitting multiple sclerosis. Mult Scler. 2005 Oct;11(5):585-91. doi: 10.1191/1352458505ms1197oa. PMID 16193898
- See also: Published in Multiple Sclerosis 2005;11:585-591 — http://www.ncbi.nlm.nih.gov/pubmed/16193898?dopt=Abstract
- See also: Full FDA approved prescribing information can be found here — http://www.mslifelines.com